CLINICAL TRIAL: NCT05820620
Title: Comparison of QLB Block and TAP Block in Terms of Pain Management and Patient Satisfaction in Morbidly Obese Patients Undergoing Laparoscopic Sleeve Gastrectomy: A Randomized Controlled Trial
Brief Title: Comparison of QLB Block and TAP Block in Morbid Obese Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biruni University (Other)
Responsible Party: Principal Investigator, Assistant Prof. Dr. Suna Koc MD, Assistant professor Dr, Biruni University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015-KAEK-76-23-02
Record Dates: First submitted 2023-03-27; First posted 2023-04-19 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Pain, Postoperative
Keywords: Morbid Obesity; TAP Block; QLB block; Analgesia
MeSH Terms: conditions — Pain, Postoperative; Obesity, Morbid; Agnosia | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: After the patients are routinely put to sleep, TAP block will be applied to the 1st group, QLB block will be applied to the 2nd group, and no intervention will be performed to the 3rd group as it is the control group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Placebo Comparator): No intervention + Patient Control Analgesia (PCA)
  Interventions: Other: Control Group
- QLB group (Experimental): QLB group Block will be applied + Patient Control Analgesia (PCA)
  Interventions: Procedure: QLB block
- TAP group (Experimental): TAP Block group will be applied + Patient Control Analgesia (PCA)
  Interventions: Procedure: TAP block

INTERVENTIONS:
Procedure: TAP block — The transversus abdominis plane (TAP) block was introduced as a landmark-guided technique via the triangle of Petit to achieve a field block. It involves the injection of a local anesthetic solution into a plane between the internal oblique muscle and transversus abdominis muscle.
  Other Names: Transversus abdominis plane (TAP)
  Arms: TAP group
Procedure: QLB block — Quadratus lumborum block is a block of the posterior abdominal wall, "interfascial plane block," which is performed exclusively under ultrasound guidance. It was described as a variant of the TAP block.
  Other Names: Quadratus lumborum block (QLB)
  Arms: QLB group
Other: Control Group — Control Group + Patient Control Analgesia (PCA)
  Arms: Control group

SUMMARY:
Quadratus lumborum block (QLB) and Transversus abdominis plane (TAP) blocks are regional anesthesia techniques that are frequently used to reduce postoperative pain and are an important part of the current analgesic regimen for many abdominal surgeries. In our clinic, researchers perform both blocks to provide postoperative analgesia. The primary aim of our study is to compare the effectiveness of TAP block and QLB block in postoperative pain control in laparoscopic sleeve gastrectomy. Secondary outcomes evaluated in this study were to assess postoperative nausea and vomiting (PONV), time to discharge, and patient satisfaction.

DETAILED DESCRIPTION:
As the number of obese patients increases, the number of surgeries performed for morbid-obese is also increasing. Pain following bariatric surgery is highly troubling and can lead to increased complication rate, decreased patient satisfaction rate, and prolonging the healing process, increasing the risk of pulmonary complications and the incidence of deep vein thrombosis. Since postoperative recovery is directly related to the severity and duration of pain, it is imperative to reduce postoperative pain as early as possible. Many post-operative methods have been suggested for patients undergoing laparoscopic surgery. Transversus abdominis plane (TAP) block is a regional anesthesia technique routinely used to reduce postoperative pain.

Quadratus lumborum block (QLB) and Transversus abdominis plane (TAP) blocks are regional anesthesia techniques that are frequently used to reduce postoperative pain and are an important part of the current analgesic regimen for many abdominal surgeries. Researchers are doing these two blocks in our clinic to provide postoperative analgesia. The aim of our study is to compare the effectiveness of TAP block and QLB block in postoperative pain control in laparoscopic sleeve gastrectomy. Secondary outcomes evaluated in this study were to assess postoperative nausea and vomiting (PONV), time to discharge, and patient satisfaction.

Many methods have been suggested to reduce postoperative abdominal wall pain, such as instillation of local anesthetics at the site of entry, patient-controlled analgesia (PCA), epidural catheterization, and the use of non-steroidal anti-inflammatory drugs (NSAIDS). It is known that opioid analgesics against acute postoperative pain cause postoperative nausea and vomiting (PONV) [3]. The mean incidence of PONV reported in the early postoperative period in patients undergoing bariatric surgery ranges from 30% to 50% [4].

Transversus abdominis plane (TAP) block is a routinely used regional anesthesia technique to reduce postoperative pain and is an important part of the current analgesic regimen for many abdominal surgeries [5]. A multimodal approach to pain management, with various combinations such as TAP blocks, local anesthetic infiltration and patient-controlled analgesia (PCA) has been suggested as the optimal combination for laparoscopic bariatric surgery [6]. Quadratus lumborum block (QLB) is one of the effective and routinely applied blocks in The primary aim of our study is to compare the effectiveness of TAP block and QLB block in postoperative pain control in laparoscopic sleeve gastrectomy. Secondary outcomes evaluated in this study were to assess postoperative nausea and vomiting (PONV), time to discharge, and patient satisfaction.

Method

Researchers planned to perform this study in a randomized controlled design in patients who will undergo laparoscopic sleeve gastrectomy in the operating room of Biruni University Hospital. After ethics committee approval, patients with BMI> 35 kg/m2, laparoscopic sleeve gastrectomy, ASA I-III, general anesthesia will be applied and patients who agree to participate in the study will be included. Patients younger than 18 years of age with bleeding disorders (INR: 1.2, antithrombotic, antiaggregant drug use, hematological disorders, etc.) that are contraindications for regional anesthesia, and those with infection at the planned skin site, psychiatric or neurological disorders, and substance addictions, will be excluded from the study.

Randomization of patients will be provided through a computer program (software). After randomization, all patients will be brought to the operating room and then put to sleep with the general anesthesia method researchers apply daily. After the patients are routinely anesthesia administration TAP block will be applied to the 1st group, QLB block will be applied to the 2nd group, and no intervention will be performed to the 3rd group as it is the control group. Blocks will be performed with 0.25% bupivacaine under USG. PCA (patient controlled analgesia) will be administered to all patients in the postoperative period to provide analgesia. For rescue analgesia; If the VAS score of the patients reaches a level of >4 and above in the postoperative period, an additional 2mg IV bolus of morphine will be administered. In cases where it is not sufficient or it is needed again, it will be intervened again with 2 mg morphine until 4 <VAS VAS score (Preop -Post op 1., 6., 12 and 24 hours) and Patient Satisfaction (Preoperative and 48 hours) (World Health Organization) WHOQOL-BREF Quality of Life Assessment and analgesic consumption amount (Morphine consumption) as evaluation parameters of the patients : Post op 1st, 6th, 12th and 24th hours). It is planned to measure the effectiveness of the blocks by measuring the pain score and patient satisfaction in the preoperative and postoperative periods, and by measuring the amount of morphine consumed (in mg). In addition, it will be checked whether there is a change in discharge times between the groups in all patients. If complications such as postoperative nausea, vomiting, allergies, nerve damage and bleeding develop, they will be recorded.

The required number of patients was determined by power analysis. In the calculation using the data of Emile et al., if 15% change is expected according to the 1st Hour VAS value of the TAP block [7]. Researchers plan a continuous study of response variables from matching study subject groups. Previous data show that the difference of matched pairs is normally distributed with a standard deviation of 1.3. If the true difference in the mean response of the matched pairs is 0.72, Researchers would need to study 28 subjects per group to reject the null hypothesis that this difference in response is zero with probability (power) 0.8. The probability of Type I error associated with this test of the 'null hypothesis' is 0.05. At least 84 patients for the three groups should be analyzed. Researchers plan to include 94 patients with a 10% probable dropout rate.

ELIGIBILITY:
Inclusion Criteria:

* BMI> 35 kg/m2
* Laparoscopic sleeve gastrectomy operation
* ASA I-III
* General anesthesia will be applied and patients who agree to participate in the study will be included.

Exclusion Criteria:

* Patients younger than 18 years of age
* Bleeding disorders (INR: 1.2, antithrombotic, antiaggregant drug use, hematological disorders, etc.) That are contraindications for regional anesthesia, and those with infection at the planned skin site
* Psychiatric or neurological disorders, and substance addictions

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2023-04-20 (Actual); Primary Completion 2024-02-20 (Actual); Study Completion 2024-02-21 (Actual)

PRIMARY OUTCOMES:
Pain management | 24th hours after surgery
  VAS value (Visual Analogue Scale) : 10cm line, with two end points representing 0 ('no pain') and 10 ('pain as bad as it could possibly be')
Pain management | 24th hours after surgery
  Morphine consumption

SECONDARY OUTCOMES:
Patient Satisfaction | Preoperative and after 7 days
  WHOQOL-BREF Quality of Life Assessment

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet I Buget, Assoc Prof, Study Director — Biruni Universty
Locations (2):
- Turkey (Türkiye) (2):
  - Suna Koç, Istanbul, Besyol
  - Suna Koç, Istanbul, Kucukcekmece

REFERENCES:
- [Result] 1. Sarandan M, Balasa CG, Papurica M et al (2011) Anesthesia in laparoscopic bariatric surgery (gastric sleeve) preliminary experience. TMJ 61:1-2
- [Result] 2. Melzack R, Katz J (1994) Pain measurements in persons in pain. In Wall PD, Melzack R (Eds) Textbook of pain. Churchill Livingstone, Edinburgh, pp 409-426
- [Result] Macintyre PE, Loadsman JA, Scott DA. Opioids, ventilation and acute pain management. Anaesth Intensive Care. 2011 Jul;39(4):545-58. doi: 10.1177/0310057X1103900405. PMID 21823370
- [Result] Sinclair DR, Chung F, Mezei G. Can postoperative nausea and vomiting be predicted? Anesthesiology. 1999 Jul;91(1):109-18. doi: 10.1097/00000542-199907000-00018. PMID 10422935
- [Result] Niraj G, Searle A, Mathews M, Misra V, Baban M, Kiani S, Wong M. Analgesic efficacy of ultrasound-guided transversus abdominis plane block in patients undergoing open appendicectomy. Br J Anaesth. 2009 Oct;103(4):601-5. doi: 10.1093/bja/aep175. Epub 2009 Jun 26. PMID 19561014
- [Result] 6. Bisgaard T (2006) Laparoskopik kolesistektomi sonrası analjezik tedavisi. Anesteziyoloji 104:835-846
- [Result] Emile SH, Abdel-Razik MA, Elbahrawy K, Elshobaky A, Shalaby M, Elbaz SA, Gado WA, Elbanna HG. Impact of Ultrasound-Guided Transversus Abdominis Plane Block on Postoperative Pain and Early Outcome After Laparoscopic Bariatric Surgery: a Randomized Double-Blinded Controlled Trial. Obes Surg. 2019 May;29(5):1534-1541. doi: 10.1007/s11695-019-03720-y. PMID 30706309